CLINICAL TRIAL: NCT01714531
Title: Improving Trauma Outcomes: A Goal Management Approach
Brief Title: Improving Outcomes After Traumatic Injury: A Goal Management Approach
Acronym: GMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristin Archer, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111484; H133G120052 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2012-10-22; First posted 2012-10-26 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Traumatic Brain Injury
Keywords: Mild TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telephone-Based Goal Management Training (Experimental): The GMT intervention targets cognitive deficits in executive functioning that impact a person's ability to carry out daily tasks. Participants learn how to recognize and stop absentmindedness and automatic pilot and how to reduce daily errors and 'slips' through goal setting. The telephone-based GMT condition includes 7 sessions delivered over the phone for 10 weeks.
  Interventions: Behavioral: Telephone-Based Goal Management Training
- Telephone-Based Attention-Control (Active Comparator): The attention group receives an educational intervention that is matched to the GMT intervention in terms of session length and contact with the study therapist. The telephone-based attention condition includes 7 sessions delivered over 10 weeks. Sessions address education on brain function and cognitive principles of memory, attention, language, perception, and motor skills. Education on stress reduction, sleep hygiene, energy management, exercise, communication, and nutrition are also provided
  Interventions: Behavioral: Telephone-Based Attention-Control
- Usual Care Control (No Intervention): Participants in the control group will receive usual care as determined by the treating surgeon. Usual care may include referral to a physical therapist, occupational therapist, psychiatrist, and/or psychologist and utilization of health services will be recorded during follow-up assessments.

INTERVENTIONS:
Behavioral: Telephone-Based Goal Management Training
  Other Names: GMT
  Arms: Telephone-Based Goal Management Training
Behavioral: Telephone-Based Attention-Control
  Arms: Telephone-Based Attention-Control

SUMMARY:
The majority of trauma survivors experience prolonged and profound physical and psychosocial disability, with up to 50% unable to return to productive employment. The Centers for Disease Control (CDC) estimates that more than 1 million of these individuals experience a mild traumatic brain injury (TBI) and cost the United States nearly $17 billion each year. Symptoms related to mild TBI result in cognitive, functional, and emotional impairments that can lead to vocational and social disability. Long-term cognitive deficits include problems with memory and attention, and most importantly executive functioning. Depressive and post-traumatic stress disorder (PTSD) symptoms are extremely common in individuals with cognitive impairment, occurring in up to 50% and 33% of individuals, respectively. The investigators have found that 55% of trauma patients with mild TBI have profound cognitive impairments in executive functioning at one-year survival. Executive functioning is defined as "a cognitive domain that controls the execution of complex activities of daily living essential for purposeful, goal directed behaviors." Deficits in executive functioning are the most disabling of all cognitive impairments and affect a person's ability to manage effectively in one's personal and professional life. Current literature shows that deficits in executive functioning contribute to reduced quality of life, difficulty in returning to work, and persistent psychological distress in various medical and surgical populations. Cognitive rehabilitation has proven effective for decreasing persistent cognitive impairment and functional disability in patients with TBI. The overall goal of cognitive rehabilitation is not only to improve a person's ability to process and interpret information but to increase self-confidence and self-efficacy for coping with emotional distress. Despite evidence supporting the use of cognitive rehabilitation, few studies have systematically addressed cognitive treatment for individuals with mild TBI. Therefore, the investigators propose to conduct a three-group randomized controlled trial to determine the efficacy of Goal Management Training (GMT), a structured manual-based intervention targeting executive functions that impact a person's ability to carry out daily tasks. The investigators hypothesize that telephone-based GMT will improve cognitive functioning, functional status, and psychological health in trauma survivors with mild TBI. Emerging research suggests that telephone rehabilitation is a feasible and effective alternative (with much broader applicability) to clinic-based interventions. Trauma survivors with mild TBI have limited access to rehabilitation services due to financial constraints and mobility and geographic restrictions that render clinic-based rehabilitation impractical. This clinical trial will recruit 90 trauma survivors with mild TBI and cognitive deficits in executive functioning. Eligible participants will be randomized to either 10-week (1) telephone-based GMT; (2) telephone-based attention-control; or (3) usual care. Primary outcomes will include observed and self-reported executive functioning and self-reported functional status as measured by a battery of standardized and previously validated cognitive tests and instruments, including the Delis-Kaplan Executive Function System Tower Test, the Dysexecutive Questionnaire, and the Functional Activities Questionnaire. Secondary outcomes will consist of depressive and PTSD symptoms, as measured by the Patient Health Questionnaire-9 and PTSD Checklist - Civilian Version, respectively. Outcome data will be collected at baseline (6 weeks after hospitalization) and at 4 month (treatment completion) and 7 month follow-up from hospital discharge. Our cognitive rehabilitation intervention will serve to broadly disseminate evidenced-based cognitive strategies to a trauma population that has difficulty returning to productive life both inside and outside the home due to profound functional and psychological disability. Findings from this study will support future research to improve the cognitive, functional and psychological health of patients following major trauma through innovative rehabilitation interventions and delivery methods.

ELIGIBILITY:
Inclusion Criteria:

1. Determination of mild TBI using American Congress of Rehabilitation Medicine guidelines;
2. No history of schizophrenia, or other psychotic disorder or suicidal intent;
3. English speaking due to feasibility of employing study personnel to deliver and assess the study intervention;
4. Age 21 years or older;
5. Able to provide a telephone number and a stable address; and
6. Presence of cognitive deficits in executive functioning (defined as 1 SD below the norm referenced mean on any 2 of the following neuropsychological tests, the D-KEF Tower Test, Trails B, and FAS)

Exclusion Criteria:

1. Having a CT scan showing an intracranial hemorrhage;
2. Current alcohol or substance abuse dependence (within the last 6 months);
3. Persons with neurological history other than TBI (e.g., premorbid epilepsy, multiple sclerosis, Alzheimer's disease);
4. Pre-existing cognitive impairment as determined by a validated surrogate or patient questionnaire (defined as a score greater than 3.3 on the IQCODE instrument;
5. History of pre-morbid learning disability;and
6. Involvement in current litigation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
D-KEFs Tower Test | 7 months after hospital discharge
  cognitive test for executive functioning
Trail Making Test B | 7 months after hospital discharge
  Cognitive test for set shifting and cognitive flexibility
Sustained Attention to Response Test | 7 months after hospital discharge
  Cognitive test for failures of sustained attention
FAS Verbal Fluency Test | 7 months after hospital discharge
  Cognitive test for verbal fluency

SECONDARY OUTCOMES:
Dysexecutive Questionnaire | 7 months after hospital discharge
  Self-reported executive functioning
Functional Activities Questionnaire | 7 months after hospital discharge
  Self-reported functional status

OTHER OUTCOMES:
Patient Health Questionnaire-9 | 7 months after hospital discharge
  Self-reported measure of depressive symptoms
PTSD Checklist-Civilian Version (PCL-C) | 7 months after hospital discharge
  Self-reported measure of PTSD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Archer, PhD, Principal Investigator — Vanderbilt School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Archer KR, Coronado RA, Haislip LR, Abraham CM, Vanston SW, Lazaro AE, Jackson JC, Ely EW, Guillamondegui OD, Obremskey WT. Telephone-based goal management training for adults with mild traumatic brain injury: study protocol for a randomized controlled trial. Trials. 2015 Jun 2;16:244. doi: 10.1186/s13063-015-0775-1. PMID 26031289